CLINICAL TRIAL: NCT05062694
Title: Physical Therapy Management Of The Patient With Central Sensitization: An Observational Study Among Italian Physiotherapists
Brief Title: Physical Therapy Management Of The Patient With Central Sensitization
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, Principal Investigator, University Hospital of Ferrara
Other Study IDs: Survey_CS
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-05

CONDITIONS: Central Sensitisation; Musculoskeletal Diseases; Pain
Keywords: Patient Management; Central Sensitisation; Muscoloskeletal Disease; Pain
MeSH Terms: conditions — Musculoskeletal Diseases; Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — It will be created a questionnaire to investigate, among Italian physiotherapists, their clinical approach to the patient with Central Sensitisation

SUMMARY:
In the literature there is still debate about the concept of central sensitization, as a pain mechanism that can support a neuromusculoskeletal pathology and which for Woolf corresponds to an amplification of neural signaling within the Central Nervous System causing hypersensitivity to pain.

This mechanism is often confused with the concept of chronic pain, as in many conditions such as fibromyalgia, traumatic neck pain, low back pain or osteoarthritis, central sensitization supports its maintenance beyond 6 months.

We believe it is important to investigate among Italian physiotherapists the management of the patient in which the presence of a central pain sensitization phenomenon is suspected, in order to provide consistent data to direct the education of health professionals towards more effective management of this problem.

To achieve this goal we aim to:

* Conduct a Delphi study in order to reach consensus, into a panel of experts, on the methods useful for the management, in each phase of the physiotherapy process, of the patient with neuromusculoskeletal problems with pain underlying central sensitization mechanism
* Investigate, through a survey among Italian physiotherapists, their clinical approach to the patient in question
* Develop a free online course available to clinical professionals and/or students who wish to deepen this issue.

ELIGIBILITY:
Inclusion Criteria:

* Italian physiotherapists who will decide to fill in the questionnaire

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physical therapists
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Physical therapists' patient management | 1 month
  Exploring Italian physiotherapists' clinical approach to the patient in question through an online survey

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria di Ferrara, Ferrara, FE, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baroni A, Margelli M, Saoncella A, Toigo I, Antonellini G, Straudi S. Physiotherapy management of nociplastic pain: A Delphi study of Italian specialists. Pain Pract. 2023 Sep;23(7):734-742. doi: 10.1111/papr.13238. Epub 2023 May 4. PMID 37143408